CLINICAL TRIAL: NCT01771250
Title: Assessment of the Effects of LY2605541 on Triglyceride Metabolism, Compared to Insulin Glargine, in Patients With Type 1 Diabetes Mellitus
Brief Title: A Study of Insulin Peglispro and Glargine on Fats in Participants With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 14871; I2R-MC-BIDN (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — basal insulin peglispro; LY2605541; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin Peglispro (Experimental): Stable dose of insulin peglispro (0.2 - 0.8 units per kilogram [U/kg]) administered subcutaneously (SC) once daily for at least 21 days in one of two treatment periods. Dose based on prestudy basal insulin dosing regimen.
  Interventions: Biological: Insulin Peglispro
- Insulin Glargine (Active Comparator): Stable dose of insulin glargine (0.2 - 0.8 U/kg) administered SC once daily for at least 21 days in one of two treatment periods. Dose based on prestudy basal insulin dosing regimen.
  Interventions: Biological: Insulin Glargine

INTERVENTIONS:
Biological: Insulin Peglispro — Daily doses administered SC.
  Other Names: LY2605541
  Arms: Insulin Peglispro
Biological: Insulin Glargine — Daily doses administered SC.
  Arms: Insulin Glargine

SUMMARY:
This study has two parts. Each participant will receive a daily injection of insulin peglispro during one treatment period and a daily injection of insulin glargine during the other treatment period. Each treatment period is 3 to 4 weeks and is followed by procedures to look at how the body uses or stores fats while taking each study drug.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetic for more than 1 year with glycated hemoglobin (HbA1c) of less than 8.5%
* Otherwise fit and healthy
* Non smoker

Exclusion Criteria:

* Taking medication or supplements other than insulin to control diabetes.
* Suffered a hypoglycemic event in the last 12 months that required hospitalization or have poor awareness of hypoglycemia
* Taking fibrates, thyroid replacement therapy, testosterone, beta blockers or systemic corticosteroids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aarhus, Denmark

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Insulin treatments were transitioned by gradual tapering/titration as required at the start of each period and the end of Period 2 based on the participants individual randomization and pre-study therapy.
Groups:
- Insulin Peglispro (LY2605541) Then Insulin Glargine: Participants took a stable dose of insulin peglispro (0.2 - 0.8 Units per kilogram [U/kg]) in Period 1 and then insulin glargine (0.2 - 0.8 U/kg) in Period 2 administered subcutaneously (SC).
- Insulin Glargine Then Insulin Peglispro: Participants took a stable dose of insulin glargine (0.2 - 0.8 U/kg) in Period 1 and then insulin peglispro (0.2 - 0.8 U/kg) in Period 2 administered subcutaneously (SC).
Period: Period 1
Arm/Group | Insulin Peglispro (LY2605541) Then Insulin Glargine | Insulin Glargine Then Insulin Peglispro
Started | 8 | 7
Received at Least One Dose of Study Drug | 7 | 7
Completed | 7 | 7
Not Completed | 1 | 0
Not completed — Met exclusion criteria | 1 | 0
Period: Period 2
Arm/Group | Insulin Peglispro (LY2605541) Then Insulin Glargine | Insulin Glargine Then Insulin Peglispro
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- All Study Participants: Participants were randomized to receive daily stable doses of either insulin peglispro or insulin glargine (0.2 -0.8 U/kg) administered SC for at least 21 days, in one of two treatment periods.
Arm/Group | All Study Participants
Number analyzed (Participants) | 14
Age, Continuous [Mean (Full Range); unit: Years] | 35.3 [22 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 14

OUTCOME MEASURES:

1. Primary Outcome: Very Low Density Lipoprotein-Triglyceride (VLDL-TG) Concentrations
Description: VLDL-TG average total concentration calculated at steady state from 240 to 420 minutes during dosing with insulin peglispro and insulin glargine.
Time Frame: Day 22: 240 minutes (min) to 420 min
Population: All participants who were randomized and received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micromole per Liter (μmol/L)
Groups:
- Insulin Peglispro: Participants took a stable dose of Insulin Peglispro (0.2 - 0.8 U/kg) administered SC once daily for at least 21 days in one of two treatment periods.
- Insulin Glargine: Participants took a stable dose of Insulin glargine (0.2 - 0.8 U/kg) administered SC once daily for at least 21 days in one of two treatment periods.
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 14 | 14
micromole per Liter (μmol/L) | 0.27 (55) | 0.17 (66)

2. Primary Outcome: VLDL-TG Secretion Rate
Description: VLDL-TG secretion rates are calculated at steady state during dosing with insulin peglispro and insulin glargine.
Time Frame: Day 22: 240 min to 420 min
Population: All participants who were randomized and took at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μmol/min
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 14 | 14
μmol/min | 38.79 (42) | 25.61 (58)

3. Primary Outcome: VLDL-TG Oxidation Rate
Description: VLDL-TG oxidation rates are calculated at steady state during dosing with insulin peglispro and insulin glargine.
Time Frame: Day 22: 240 min to 420 min
Population: All participants who were randomized and received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μmol/min
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 14 | 14
μmol/min | 20.13 (40) | 15.34 (59)

4. Primary Outcome: VLDL-TG Clearance Rate
Description: VLDL-TG clearance rates are calculated at steady state during dosing with insulin peglispro and insulin glargine.
Time Frame: Day 22: 240 min to 420 min
Population: All participants who were randomized and received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliters per minute (mL/min)
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 14 | 14
milliliters per minute (mL/min) | 142.16 (47) | 155.11 (49)

ADVERSE EVENTS:
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Insulin Peglispro | Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 0/14 | 1/14
Other Adverse Events (participants affected / at risk) | 4/14 | 5/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Peglispro (N=14) | Insulin Glargine (N=14)
Dermoid cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Peglispro (N=14) | Insulin Glargine (N=14)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No